CLINICAL TRIAL: NCT00027820
Title: Low-Dose TBI and Fludarabine Followed by Nonmyeloablative Unrelated Donor Peripheral Blood Stem Cell Transplantation Using Enhanced Postgrafting Immunosuppression for Patients With Hematologic Malignancies and Renal Cell Carcinoma - A Multi-center Trial
Brief Title: Total-Body Irradiation and Fludarabine Phosphate Followed by Donor Peripheral Blood Stem Cell Transplant in Treating Patients With Hematologic Malignancies or Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1641.00; NCI-2012-00591 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1641.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01CA018029 (NIH)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Myelodysplastic Syndrome; Childhood Renal Cell Carcinoma; Chronic Myelomonocytic Leukemia; Clear Cell Renal Cell Carcinoma; de Novo Myelodysplastic Syndrome; Metastatic Renal Cell Cancer; Previously Treated Myelodysplastic Syndrome; Progression of Multiple Myeloma or Plasma Cell Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult Non-Hodgkin Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Non-Hodgkin Lymphoma; Refractory Anemia; Refractory Anemia With Ringed Sideroblasts; Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Renal Medullary Carcinoma; Type 1 Papillary Renal Cell Carcinoma; Type 2 Papillary Renal Cell Carcinoma; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia; Untreated Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Carcinoma, Renal Cell; Leukemia, Plasma Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Hodgkin Disease; Lymphoma, Non-Hodgkin; Anemia, Refractory; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine phosphate; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Cyclosporine; Cyclosporins; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (PBSCT) (Experimental): REDUCED-INTENSITY CONDITIONING: Patients receive fludarabine phosphate IV on days -4, -3, and -2 and undergo TBI on day 0.
  TRANSPLANT: Patients undergo allogeneic PBSCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID on days -3 to 100 with taper to day 177 and mycophenolate mofetil PO every 8 hours on days 0-40 with taper to day 96.
  Interventions: Drug: Fludarabine Phosphate; Radiation: Total-Body Irradiation; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; SH T 586
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; Total Body Irradiation; Whole-Body Irradiation
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo nonmyeloablative PBSCT
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo nonmyeloablative PBSCT
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Drug: Cyclosporine — Given PO
  Other Names: 27-400; CsA; Neoral; OL 27-400; Sandimmun
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF

SUMMARY:
This phase I/II trial studies whether a new kind of blood stem cell (bone marrow) transplant, that may be less toxic, is able to treat underlying blood cancer. Stem cells are "seed cells" necessary to make blood cells. Researchers want to see if using less radiation and less chemotherapy with new immune suppressing drugs will enable a stem cell transplant to work. Researchers are hoping to see a mixture of recipient and donor stem cells after transplant. This mixture of donor and recipient stem cells is called "mixed-chimerism". Researchers hope to see these donor cells eliminate tumor cells. This is called a "graft-versus-leukemia" response.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether stable unrelated peripheral blood stem cell (PBSC) grafts can be safely established using nonmyeloablative pretransplant conditioning with intensified post-grafting immunosuppression and with every (q) 8 hours (hr) and possibly q 6 hr mycophenolate mofetil (MMF) dosing in patients with hematologic malignancies and renal cell carcinoma.

II. To determine if the incidence and severity of acute grades II-IV graft-versus-host disease (GVHD) can be reduced in patients with sustained engraftment with the use of q 8 hr MMF dosing.

SECONDARY OBJECTIVES:

I. To determine if engraftment can be maintained in patients with low chimerism and high risk of rejection with the use of a single dose of fludarabine (fludarabine phosphate) followed by donor lymphocyte infusion (DLI) on continued MMF/cyclosporine (CSP).

II. To compare survival and disease free survival to those achieved under protocol 1463.

OUTLINE:

REDUCED-INTENSITY CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) on days -4, -3, and -2 and undergo total-body irradiation (TBI) on day 0.

TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell transplant (PBSCT) on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) twice daily (BID) on days -3 to 100 with taper to day 177 and mycophenolate mofetil PO every 8 hours on days 0-40 with taper to day 96.

After completion of study treatment, patients are followed up at 6 months, 1 year, 1.5 years, 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 50 years with hematologic malignancies treatable by unrelated hematopoietic stem cell transplantation (HSCT)
* Ages =< 50 years of age with hematologic diseases treatable by allogeneic HSCT who through pre-existing medical conditions or prior therapy are considered to be at high risk for regimen related toxicity associated with a conventional transplant (> 40% risk of transplant related mortality [TRM]) or those patients who refuse a conventional HSCT; transplants must be approved for these inclusion criteria by both the participating institution's patient review committee such as the Patient Care Conference (PCC at the Fred Hutchinson Cancer Research Center [FHCRC]) and by the principal investigator at the collaborating center; patients =< 50 years of age who have received previous autologous transplantation do not require patient review committee approval; all children < 12 years must be discussed with the FHCRC principal investigator (PI) prior to registration
* Patients with metastatic renal cell carcinoma with the histologic subtypes of clear cell, papillary and medullary may be accepted regardless of age
* The following diseases will be permitted although other diagnoses can be considered if approved by PCC or the participating institution's patient review committees and the principal investigator:

  * Intermediate or high grade non-Hodgkin lymphoma (NHL) - not eligible for autologous HSCT or after failed autologous HSCT
  * Low grade NHL - with < 6 month duration of complete remission (CR) between courses of conventional therapy
  * Chronic lymphocytic leukemia (CLL) - must have failed two lines of conventional therapy and be refractory to fludarabine
  * Hodgkin's disease (HD) - must have received and failed frontline therapy
  * Multiple myeloma (MM) - must have received prior chemotherapy; consolidation of chemotherapy by autografting prior to nonmyeloablative HSCT is permitted
  * Acute myeloid leukemia (AML) - must have < 5% marrow blasts at the time of transplant
  * Acute lymphoblastic leukemia - must have < 5% blasts at the time of transplant
  * Chronic myelogenous leukemia (CML) - patients will be accepted in chronic phase or accelerated phase; patients who have received prior autografts after high dose therapy or have undergone intensive chemotherapy with PBSC autologous or conventional HSCT for advanced CML may be enrolled provided they are in CR or chronic phase (CP) and have < 5% marrow blasts at time of transplant
  * Myelodysplastic syndromes (MDS)/myeloproliferative disorder (MPD) - only patients with MDS/refractory anemia (RA) or MDS/refractory anemia with ringed sideroblasts (RARS) will be eligible for this protocol; additionally patients with myeloproliferative syndromes (MPS) will be eligible; those patients with MDS or MPS with > 5% marrow blasts (including those with transformation to AML) must receive cytotoxic chemotherapy and achieve < 5% marrow blasts at time of transplant
  * Renal cell carcinoma - must have evidence of disease not amenable to surgical cure or history of or active metastatic disease by radiological and histologic criteria
* DONOR: FHCRC matching allowed will be grade 1.0 to 2.1; unrelated donors who are prospectively:

  * Matched for human leukocyte antigen (HLA)-A, B, C, DRB1 and DQB1 by high resolution typing
  * Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* DONOR: A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
* DONOR: Patient and donor pairs homozygous at a mismatched allele are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0201, and this type of mismatch is not allowed
* DONOR: PBSC only will be permitted as a hematopoietic stem cell (HSC) source on this protocol

Exclusion Criteria:

* Patients with rapidly progressive intermediate or high grade NHL
* Renal cell carcinoma patients:

  * With expected survival of less than 6 months
  * Disease resulting in severely limited performance status (< 70%)
  * Any vertebral instability
  * History of brain metastases
* Central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant
* Patients with non-hematological tumors except renal cell carcinoma
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Cardiac ejection fraction < 35%; ejection fraction is required if there is a history of anthracycline exposure or history of cardiac disease
* Diffusion capacity of the lung for carbon monoxide (DLCO) < 40% and/or receiving supplementary continuous oxygen
* The FHCRC PI of the study must approve of enrollment of all patients with pulmonary nodules
* Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease
* Karnofsky scores < 60 (except renal cell carcinoma [RCC])
* Patients with > grade II hypertension by common toxicity criteria (CTC)
* Human immunodeficiency virus (HIV) positive patients
* The addition of cytotoxic agents for "cytoreduction" with the exception of hydroxyurea and imatinib mesylate will not be allowed within two weeks of the initiation of conditioning
* DONOR: Marrow donors
* DONOR: Donors who are HIV-positive and/or, medical conditions that would result in increased risk for filgrastim (G-CSF) mobilization and harvest of PBSC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2001-08; Primary Completion 2004-09 (Actual); Study Completion 2004-09-05 (Actual)

PRIMARY OUTCOMES:
Risk of true graft rejection in patients with and without preceding chemotherapy | Up to 5 years
  The goal is to reduce the risk in patients without preceding chemotherapy to < 20% and with preceding chemotherapy to < 10%.
Risk of grades II-IV acute GVHD in those patients with sustained engraftment | Up to 5 years
  The goal is to reduce the incidence of grades II-IV acute GVHD from 50% to less than 35% in patients with sustained engraftment by increasing the dosing of MMF to every 8 hours. The impact of the enhanced post-grafting immunosuppression on objective measures of GVHD will be described. These include doses and duration of immunosuppression (in particular corticosteroids) and number of GVHD treatment regimens used within the first year. These parameters will be compared to the results of protocol 1463.

SECONDARY OUTCOMES:
Incidence of reversing impending graft rejection (less than 40% donor cluster of differentiation [CD]3+ T cell chimerism) | Up to 5 years
  The secondary objective of reversing pending graft rejection with fludarabine phosphate and DLI will be evaluated in the context of overall engraftment. The number of patients given DLI in this context is expected to be small. The response to DLI will be followed and reported in a descriptive manner. The effect of this intervention on adverse outcomes will be followed.
Overall survival | Up to 5 years
Progression-free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (10):
- United States (8):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Stanford University Hospitals and Clinics, Stanford, California
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Baylor Medical Center at Garland, Garland, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Universitaet Leipzig, Leipzig, Germany
- University of Torino, Torino, Italy

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241